CLINICAL TRIAL: NCT02509052
Title: A Phase I/II Dose-Escalation Trial of Leflunomide in Patients With Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Leflunomide in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15140; NCI-2015-01181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15140 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Leflunomide

STUDY DESIGN:
Intervention Model Description: The phase I portion will implement a modified rolling six dose escalation design, a more conservative version of the rolling six design of Skolnik, et al., for enrollment with dose escalation, de-escalation, or expansion of a cohort on the basis of the occurrence of dose limiting toxicities (DLTs) during cycle 1. The starting dose of leflunomide is 20mg daily, with the intention to test up to 60mg daily. Escalation will proceed in increments of 20mg/daily; de-escalation will proceed in decrements of 10mg/day. Leglunomide is administered with a loading dose of 100 mg for the 1st three doses.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: 20 mg leflunomide (Experimental): Patients receive 20 mg leflunomide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Leflunomide; Other: Pharmacological Study
- Arm 2: 40 mg leflunomide (Experimental): Patients receive 40 mg leflunomide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Leflunomide; Other: Pharmacological Study
- Arm 3: 60 mg leflunomide (Experimental): Patients receive 60 mg leflunomide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Leflunomide; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leflunomide — Given PO
  Other Names: Arava; SU101
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of leflunomide in treating patients with multiple myeloma that has come back (relapsed) or has not responded to previous treatment (refractory). Leflunomide may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of leflunomide, when given as a single agent. (Phase I) II. To assess the safety and tolerability of leflunomide at each dose level by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration. (Phase I) III. To evaluate the anti-myeloma activity of leflunomide, when given as a single agent, as assessed by overall response rate (ORR). (Phase II)

SECONDARY OBJECTIVES: I. To obtain estimates of: response duration, clinical benefit response, overall survival, progression-free survival. (Phase II)

TERTIARY OBJECTIVES: I. To characterize the relationship between serum concentration of the active leflunomide metabolite, teriflunomide (A77 1726), and toxicity. (Phase I/II) II. To assess the relationship between serum concentration of the active leflunomide metabolite, teriflunomide (A77 1726), and disease response. (Phase I/II) III. To explore the relationship between polymorphisms in the CYP1A2, CYP2C19, or DHODH genes and toxicity/response. (Phase I/II) IV. To explore the ex vivo cytotoxicity of leflunomide toward primary multiple myeloma (MM) cells, in order to evaluate whether individual ex vivo leflunomide response might be a useful predictor of therapeutic response. (Phase I/II) V. To explore the potential additive or synergistic effects of combining leflunomide with other classes of Food and Drug Administration (FDA)-approved drugs. (Phase I/II) VI. To generate a preliminary ribonucleic acid (RNA)/microRNA (miRNA) and deoxyribonucleic acid (DNA) methylation signature associated with response of MM cells to leflunomide in vivo (mRNA/miRNA and DNA methylation, phase II only) and teriflunomide ex vivo (messenger RNA [mRNA]/miRNA). (Phase I/II)

OUTLINE: This is a dose-escalation study. Patients receive leflunomide orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up at 30 days and then every 28 days until disease progression (active follow-up) or every 3 months (long term follow-up).

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients must have a life expectancy of > 3 months
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must have a diagnosis of multiple myeloma
* Serum M-protein >= 0.5 g/dL
* Urine M-protein >= 200 mg/24 hr
* Serum free light chain >=10 mg/dL provided the free light chain (FLC) ratio is abnormal
* 10% plasma cells in bone marrow
* Patients must be relapsed or are refractory to at least 3 prior lines of therapy, including both a proteasome inhibitor an immunomodulatory drug (IMiD), and for whom a transplant is not recommended (induction therapy and stem cell transplant +/- maintenance will be considered as one regimen)
* At least 2 weeks from prior therapy to time of start of treatment; prior therapy includes steroids (except prednisone or equivalent - up to 10 mg per day is allowed)
* Platelet count >= 50,000/uL; platelet transfusions are not allowed within 14 days of platelet assessment
* Absolute neutrophil count (ANC) >= 1000/mm^3; growth factor is not permitted within 14 days of neutrophil assessment
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.0 x upper limit of normal (ULN)
* Total Bilirubin < 1.5 x ULN
* Calculated creatinine clearance (CrCl) >= 30 mL/min per 24 hour urine collection or the Cockcroft-Gault formula
* Negative serum or urine beta-human chorionic gonadotropin (B-HCG) test (female patient of childbearing potential* only), to be performed locally within the screening period
* Negative for tuberculosis antigen (e.g. T-Spot test)
* Negative for hepatitis A, B, or C infection
* Adequate pulmonary function as defined by forced vital capacity (FVC) and diffusing capacity of the lung for carbon monoxide (DLCO) >= 50% of predicted by pulmonary function testing
* Agreement by females of childbearing potential* and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for three months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately * A female of childbearing potential is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months

Exclusion Criteria:

* Prior treatment with leflunomide
* Current or planned use of other investigational agents, or concurrent biological, chemotherapy, or radiation therapy during the study treatment period
* Current or planned growth factor or transfusion support until after initiation of treatment; if growth factor or transfusion support is provided between screening and start of treatment, the participant will no longer be eligible
* Prior diagnosis of rheumatoid arthritis
* Prior allogenic transplant
* Acute active infection requiring systemic therapy within 2 weeks prior to enrollment
* Pre-existing liver disease
* Known human immunodeficiency virus (HIV) infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to leflunomide or cholestyramine
* Non-hematologic malignancy within the past 3 years aside from the following exceptions:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Prostate cancer < Gleason grade 6 with a stable prostate specific antigen (PSA)
  * Successfully treated in situ carcinoma of the breast
* Clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or the patient's ability to give informed consent
* Pregnant women and women who are lactating; breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc
* NONCOMPLIANCE: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosenzweig, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Rosenzweig M, Palmer J, Tsai NC, Synold T, Wu X, Tao S, Hammond SN, Buettner R, Duarte L, Htut M, Karanes C, Nathwani N, Pichiorri F, Sahebi F, Sanchez JF, Chowdhury A, Krishnan A, Forman SJ, Rosen ST. Repurposing leflunomide for relapsed/refractory multiple myeloma: a phase 1 study. Leuk Lymphoma. 2020 Jul;61(7):1669-1677. doi: 10.1080/10428194.2020.1742900. Epub 2020 Apr 8. PMID 32268821

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol was formerly designed as a Phase I/II trial. New preclinical trial data were cause for us to conclude the trial before beginning the phase II portion.
Period: Overall Study
Arm/Group | Arm 1: 20 mg Leflunomide | Arm 2: 40 mg Leflunomide | Arm 3: 60 mg Leflunomide
Started | 3 | 3 | 6
Completed | 3 | 3 | 5
Not Completed | 0 | 0 | 1
Not completed — Non compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Because we obtained preclinical data indicating a synergistic effect between leflunomide and lenalidomide, we determined that investigating leflunomide-based combinational therapy was favorable over pursuing a phase 2 study of single-agent leflunomide. There were no dose de-escalations, so there were no patients accrued to the arms for 10mg, 30mg, or 50mg.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 20 mg Leflunomide | Arm 2: 40 mg Leflunomide | Arm 3: 60 mg Leflunomide | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Continuous [Median (Full Range); unit: years] | 50 [48 to 72] | 62 [60 to 67] | 71 [64 to 85] | 68 [48 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 6
  Male | 2 | 2 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race/ethnicity: Asian | 0 | 1 | 1 | 2
  race/ethnicity: Black | 2 | 1 | 1 | 4
  race/ethnicity: Hispanic or Latino | 0 | 1 | 0 | 1
  race/ethnicity: White, non-Hispanic | 1 | 0 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 12
ISS staging at diagnosis [Count of Participants; unit: Participants] — The International Staging System (ISS) consists of the following stages:
  Stage I - serum beta-2 microglobulin less than 3.5 mg/L AND serum albumin greater than or equal to 3.5 g/dL ::
  Stage II - neither stage I nor III ::
  stage III - serum beta-2 microglobulin greater than or equal to 5.5 mg/L :: Higher grade predicts worse outcome.
  J Clin Oncol 23:3412-3420
  Participants
    Stage I | 2 | 1 | 0 | 3
    Stage II | 0 | 1 | 2 | 3
    Stage III | 0 | 1 | 2 | 3
    Unknown/missing | 1 | 0 | 2 | 3
Prior autologous transplant [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 4 | 10
  No | 0 | 0 | 2 | 2
Prior radiation [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 1 | 4
  No | 2 | 1 | 5 | 8
Serum electrophoresis and immunofixation [Count of Participants; unit: Participants] — Serum protein electrophoresis refers to the separation of different types of proteins, according to the differences in the surface charge of serum proteins. Immunoglobulin (Ig) exhibits tetrapeptide chain structure, which can be divided into five categories: IgA, IgM, IgD, IgE, or IgG. Serum Ig can be used in diagnosis of MM. Immunofixation electrophoresis involves the dissociation of electrophoresis and the high specificity (antigen-antibody reaction) and high sensitivity of monoclonal immunoglobulin to detect monoclonal components in serum. J Coll Physicians Surg Pak 2021; 31(07):864-867
  Participants
    Positive | 2 | 3 | 6 | 11
    Negative | 1 | 0 | 0 | 1
Type of positive serum electrophoresis and immunofixation patients [Count of Participants; unit: Participants] — Serum protein electrophoresis refers to the separation of different types of proteins, according to the differences in the surface charge of serum proteins. Immunoglobulin (Ig) exhibits tetrapeptide chain structure, which can be divided into five categories: IgA, IgM, IgD, IgE, or IgG. Serum Ig can be used in diagnosis of MM. Immunofixation electrophoresis involves the dissociation of electrophoresis and the high specificity (antigen-antibody reaction) and high sensitivity of monoclonal immunoglobulin to detect monoclonal components in serum. J Coll Physicians Surg Pak 2021; 31(07):864-867 Population: This is division of the Positive patients.
  Participants
    IgG kappa | 1 | 1 | 3 | 5
    IgG lambda | 0 | 1 | 2 | 3
    IgA lambda | 0 | 0 | 0 | 0
    Serum unknown | 1 | 0 | 1 | 2
    IgA kappa | 1 | 1 | 0 | 2
PI refractory [Count of Participants; unit: Participants] — PI (proteasome inhibitor) refractory is disease that is non-responsive to therapy with bortezomib, or progressing within 60 days of cessation of the most recent bortezomib therapy in patients who have achieved minimal response (MR) or better.
  Participants
    Yes | 3 | 3 | 4 | 10
    No | 0 | 0 | 2 | 2
IMiD refractory [Count of Participants; unit: Participants] — IMiD (immunomodulatory drug) refractory is disease that is non-responsive to therapy with lenalidomid, or progressing within 60 days of cessation of the most recent lenalidomid therapy in patients who have achieved minimal response (MR) or better.
  Participants
    Yes | 1 | 3 | 6 | 10
    No | 2 | 0 | 0 | 2
Double refractory (bortezomib/lenalidomide) [Count of Participants; unit: Participants] — Double refractory is disease that is non-responsive to therapy with either bortezomib or lenalidomide, or progressing within 60 days of cessation of the most recent therapy with either bortezomib or lenalidomide in patients who have achieved minimal response (MR) or better.
  Participants
    Yes | 1 | 3 | 4 | 8
    No | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: MTD, Defined as the Highest Dose in Which =< 1/6 Patients Experience a Dose-limiting Toxicity, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03
Description: Observed toxicities will be summarized, for all dose levels, in terms of type (organ affected or laboratory determination), severity, time of onset, duration, serum concentration of the active leflunomide metabolite, probable association with the study treatment and reversibility or outcome.
Time Frame: 28 days
Population: Recommended phase 2 dose: This was the highest planned dose level within this study. Because we obtained preclinical data indicating a synergistic effect between leflunomide and lenalidomide, we determined that investigating leflunomide-based combinational therapy was favorable over pursuing a phase 2 study of single-agent leflunomide. There were no dose de-escalations, so there were no patients accrued to the arms for 10mg, 30mg, or 50mg.
Measure: Number; unit: mg
Groups:
- All Participants: Patients receive 20, 40 or 60 mg leflunomide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Participants
Number analyzed (Participants) | 12
mg | 60

2. Primary Outcome: Best Overall Response Rate: Proportion of Patients Reaching CR by IMWG Criteria
Description: Stringent complete response [sCR]/complete response [CR]/very good partial response [VGPR]/or partial response [PR]), assessed by International Myeloma Working Group (IMWG) criteria.
Time Frame: From the start of treatment until disease progression/recurrence, assessed up to 48 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 20 mg Leflunomide | Arm 2: 40 mg Leflunomide | Arm 3: 60 mg Leflunomide
Number analyzed (Participants) | 3 | 3 | 5
Participants | 3 | 3 | 3

3. Secondary Outcome: Clinical Benefit Response Rate (sCR/CR/VGPR/Partial Response [PR]/Minimal Response [MR] or Stable Disease [SD]), Assessed by IMWG Criteria
Description: Clinical benefit response rate (sCR/CR/VGPR/partial response [PR]/minimal response [MR] or stable disease [SD]), assessed by International Myeloma Working Group (IMWG) criteria
Time Frame: From the start of treatment until disease progression/recurrence, assessed up to 48 months
Population: Evaluable patients. One patient was non-compliant, therefore, inevaluable. Because we obtained preclinical data indicating a synergistic effect between leflunomide and lenalidomide, we determined that investigating leflunomide-based combinational therapy was favorable over pursuing a phase 2 study of single-agent leflunomide. There were no dose de-escalations, so there were no patients accrued to the arms for 10mg, 30mg, or 50mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 20 mg Leflunomide | Arm 2: 40 mg Leflunomide | Arm 3: 60 mg Leflunomide
Number analyzed (Participants) | 3 | 3 | 5
Participants | 3 | 3 | 3

4. Secondary Outcome: Response Duration
Description: Median and range of nine patients with Complete Response (CR)
Time Frame: Assessed up to 48 months
Population: Among the 12 enrolled patients, only 11 patients are evaluable for response. And 9 of the 11 evaluable patients reached CR. The response duration is based on these 9 CR patients.
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: 20 mg Leflunomide | Arm 2: 40 mg Leflunomide | Arm 3: 60 mg Leflunomide
Number analyzed (Participants) | 3 | 3 | 3
days | 336 [28 to 401] | 112 [91 to 152] | 54 [28 to 56]

5. Secondary Outcome: Response Duration
Description: Number of patients with Stable Disease greater than or equal to 90 days
Time Frame: Assessed at ninety days.
Population: Nine patients who reached CR among 11 patients evaluable for response. Because we obtained preclinical data indicating a synergistic effect between leflunomide and lenalidomide, we determined that investigating leflunomide-based combinational therapy was favorable over pursuing a phase 2 study of single-agent leflunomide. There were no dose de-escalations, so there were no patients accrued to the arms for 10mg, 30mg, or 50mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 20 mg Leflunomide | Arm 2: 40 mg Leflunomide | Arm 3: 60 mg Leflunomide
Number analyzed (Participants) | 3 | 3 | 3
Participants | 2 | 3 | 0

ADVERSE EVENTS:
Time Frame: up to thirty days post-treatment.
Arm/Group | Arm 1: 20 mg Leflunomide | Arm 2: 40 mg Leflunomide | Arm 3: 60 mg Leflunomide
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/3 | 2/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 4/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: 20 mg Leflunomide (N=3) | Arm 2: 40 mg Leflunomide (N=3) | Arm 3: 60 mg Leflunomide (N=6)
10016558-Fever (General disorders) | 1 | 0 | 0
10040047-Sepsis (Infections and infestations) | 0 | 0 | 1
10046571-Urinary tract infection (Infections and infestations) | 0 | 0 | 1
10061229-Lung infection (Infections and infestations) | 0 | 1 | 1
10017076-Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
10003481-Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
10023838-Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: 20 mg Leflunomide (N=3) | Arm 2: 40 mg Leflunomide (N=3) | Arm 3: 60 mg Leflunomide (N=6)
10002272-Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0
10025182-Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1
10033557-Palpitations (Cardiac disorders) | 0 | 0 | 1
10040752-Sinus tachycardia (Cardiac disorders) | 1 | 0 | 3
10061389-Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 1
10061589-Aortic valve disease (Cardiac disorders) | 0 | 0 | 1
10014020-Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
10005886-Blurred vision (Eye disorders) | 0 | 1 | 0
10034960-Photophobia (Eye disorders) | 0 | 0 | 1
10000081-Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
10008417-Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
10010774-Constipation (Gastrointestinal disorders) | 0 | 2 | 1
10012727-Diarrhea (Gastrointestinal disorders) | 2 | 2 | 2
10028813-Nausea (Gastrointestinal disorders) | 1 | 2 | 2
10044055-Toothache (Gastrointestinal disorders) | 0 | 1 | 0
10047700-Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
10008531-Chills (General disorders) | 1 | 0 | 2
10014222-Edema face (General disorders) | 1 | 0 | 0
10016059-Facial pain (General disorders) | 1 | 0 | 0
10016256-Fatigue (General disorders) | 2 | 3 | 4
10016558-Fever (General disorders) | 0 | 0 | 3
10017577-Gait disturbance (General disorders) | 0 | 1 | 0
10025482-Malaise (General disorders) | 0 | 0 | 1
10033371-Pain (General disorders) | 0 | 2 | 3
10054482-Neck edema (General disorders) | 1 | 0 | 0
10062466-Localized edema (General disorders) | 1 | 0 | 1
10062501-Non-cardiac chest pain (General disorders) | 1 | 0 | 0
10040872-Skin infection (Infections and infestations) | 1 | 0 | 0
10046300-Upper respiratory infection (Infections and infestations) | 1 | 1 | 0
10046571-Urinary tract infection (Infections and infestations) | 0 | 0 | 3
10016173-Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
10001551-Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
10003481-Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
10005364-Blood bilirubin increased (Investigations) | 1 | 0 | 1
10011368-Creatinine increased (Investigations) | 0 | 2 | 1
10025256-Lymphocyte count decreased (Investigations) | 1 | 1 | 1
10029366-Neutrophil count decreased (Investigations) | 3 | 3 | 2
10035528-Platelet count decreased (Investigations) | 2 | 3 | 5
10047896-Weight gain (Investigations) | 0 | 0 | 1
10047900-Weight loss (Investigations) | 1 | 1 | 2
10049182-White blood cell decreased (Investigations) | 3 | 3 | 2
10002646-Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 4
10012174-Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
10020587-Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
10020670-Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
10020870-Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 1
10020907-Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 3
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2
10021005-Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2 | 2
10021018-Hypokalemia (Metabolism and nutrition disorders) | 0 | 3 | 3
10021028-Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
10021038-Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 3
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0
10003239-Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
10006002-Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
10016750-Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
10028836-Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
10033425-Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
10039722-Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
10062572-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
10029104-Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
10013573-Dizziness (Nervous system disorders) | 0 | 1 | 2
10019211-Headache (Nervous system disorders) | 1 | 1 | 1
10041349-Somnolence (Nervous system disorders) | 0 | 0 | 1
10002855-Anxiety (Psychiatric disorders) | 0 | 0 | 1
10010300-Confusion (Psychiatric disorders) | 0 | 0 | 2
10022437-Insomnia (Psychiatric disorders) | 1 | 0 | 2
10019450-Hematuria (Renal and urinary disorders) | 0 | 0 | 2
10037032-Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
10046539-Urinary frequency (Renal and urinary disorders) | 0 | 0 | 2
10046912-Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
10001723-Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
10028735-Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
10035623-Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
10037400-Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
10038738-Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
10041367-Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
10020642-Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
10020407-Hot flashes (Vascular disorders) | 1 | 0 | 0
10020772-Hypertension (Vascular disorders) | 3 | 2 | 5
10021097-Hypotension (Vascular disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT02509052/Prot_SAP_000.pdf